CLINICAL TRIAL: NCT04975178
Title: Randomised, Double-Blind, Controlled Phase 3 Trial to Evaluate the Efficacy, Safety and Immunogenicity of MTBVAC in Healthy HIV Unexposed (HU) and HIV Exposed Uninfected (HEU) Newborns in Tuberculosis-Endemic Regions of Sub-Saharan Africa
Brief Title: Efficacy, Safety and Immunogenicity Evaluation of MTBVAC in Newborns in Sub-Saharan Africa
Acronym: MTBVACN3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biofabri, S.L (Industry)
Collaborators: TuBerculosis Vaccine Initiative (Other); University of Cape Town (Other); Institut Pasteur de Madagascar (Other); Biomedical Research Center EPLS (Other); Universidad de Zaragoza (Other); University of Stellenbosch (Other); University of KwaZulu (Other); Wits Health Consortium (Pty) Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTBVACN3
Record Dates: First submitted 2021-06-21; First posted 2021-07-23 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — MTBVAC vaccine

STUDY DESIGN:
Intervention Model Description: The study is designed to include the following:
  1. Safety population (all study participants randomized to receive BCG or MTBVAC in a 1:1 fashion): All participants from the 4 South African sites (approx. 7000); all 120 participants from Madagascar & Senegal.
  2. Reactogenicity population:
     - First 1000 from the 4 South African sites and all 120 in Madagascar and Senegal.
  3. Immunogenicity population (subset of the safety population - total 460):
     - First 60 HU and 25 HEU participants from the South African sites (total 340) and all 120 from Madagascar & Senegal.
  4. Efficacy population (subset of the safety population - all participants from the South African sites):
     * First 1000, including 240 HU and 100 HEU newborns.
     * Additional 6000 (not part of reactogenicity & immunogenicity population). Senegal & Madagascar participants are excluded from the efficacy population. DSMB will periodically review cumulative safety and reactogenicity data.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: MTBVAC and BCG vaccine will be prepared, and allocation concealed by the site pharmacist. All other site staff will be blinded to vaccine allocation, throughout the follow-up period. Data pertaining to the MTBVAC vaccine and to BCG control will be collected in an observer-blinded manner. Blinding will be maintained throughout the vaccination and follow-up portions of the vaccine trial. No set of individual codes will be held at Biofabri's Headquarters. Biofabri's Headquarters will be able to access the individual randomization code from the SATVI Pharmacy randomization register. The code will be broken by the Site's Pharmacist (Study Contact for Emergency Code Break) only in the case of medical events that the investigator/physician in charge of the participant feels cannot be treated without knowing the identity of the study vaccine(s). The Site's Pharmacist is responsible for unblinding the treatment assignment in accordance with specified time frames for expedited reporting of SAEs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MTBVAC (Experimental): Both MTBVAC and BCG vaccines are administered by intradermal route in the left deltoid region. One 0.05 mL reconstituted dose of MTBVAC will be defined based on the phase IIa results.
  MTBVAC is manufactured by Biofabri. MTBVAC is formulated (1.5 - 8.5 x104 CFU/dose, 1.5 - 8.5 x105 CFU/dose or 1.5 - 8.5 x106 CFU/dose (to be selected) and presented as a lyophilised pellet in 20 dose vials (0.05 mL/dose, after reconstitution with sterile water for injection). MTBVAC vaccine will be released and distributed by BIOFABRI, and imported to the sites following approval by the local regulatory authority. MTBVAC vaccine must be stored at +2°C to +8°C. Reconstituted MTBVAC vaccine must be stored at +2ºC to +8ºC and administered as soon as possible, within 4 hours of reconstitution. A single vaccine vial will be used for each participant.
  Interventions: Biological: MTBVAC
- BCG (Active Comparator): BCG is a live attenuated M. bovis strain developed 100 years ago and is used as a preventive vaccine against tuberculosis. It is administered at birth.
  One 0.05 mL reconstituted dose of BCG contains 2.5 x 105 CFU. The control vaccine will be the BCG vaccine available and recommended in South Africa at time of the trial.
  BCG vaccine produced by AJ Biologics (formerly Staten Serum Institute) is the only BCG vaccine (Danish strain) currently licensed for routine use in South Africa. The recommended BCG injection volume for newborn infants (0.05 mL, after reconstitution with BCG diluent) contains approximately 2.5 x 105 CFU (range 1-4 x 105 CFU). BCG vaccine vials should be stored in the site pharmacy at 2-8ºC.
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: MTBVAC — MTBVAC is a novel TB vaccine candidate based on an attenuated M. tuberculosis clinical isolate of the Euro-American lineage. Attenuation is based on two independent, stable genetic deletions of the genes phoP and fadD26 coding for two major virulence factors, the transcription factor PhoP and the cell-wall lipids PDIM, respectively. We hypothesize that MTBVAC will provide improved protection, as individuals latently infected with live M.tuberculosis have an 80% lower chance of developing TB, and as MTBVAC contains most of the genes deleted from BCG and presents a wider collection of antigens to the host immune system. Preclinical studies in different animal models indicated that MTBVAC is safe and is able to induce an improved protection compared to BCG.
  Arms: MTBVAC
Biological: BCG — BCG is a live attenuated M. bovis strain developed 100 years ago and is used as a preventive vaccine against tuberculosis. It is administered at birth.
  Arms: BCG

SUMMARY:
The objective of this project is to demonstrate safety, immunogenicity and improved efficacy of the new live attenuated M. tuberculosis vaccine called MTBVAC in a Phase 3 efficacy trial in HIV-uninfected infants born to HIV-infected and HIV-uninfected mothers as compared to standard of care BCG vaccination. The proposal builds upon a group of TB vaccine development partners in Europe and sub-Saharan Africa established in a previous EDCTP-supported project. It creates an expanded consortium of clinical trial partners for the optimal implementation of a large infant efficacy trial of MTBVAC in high TB incidence settings. New capacity for efficacy trials in infants will be a valuable resource for the TB vaccine development community. The proposal will create a network of institutions in three TB endemic African countries with enhanced laboratory capacity to conduct TB vaccine immunology studies and to bio-bank samples to discover immune correlates of vaccine-mediated protection.

DETAILED DESCRIPTION:
A new effective tuberculosis (TB) vaccine is essential to achieve World Health Organization End TB goals and eliminate TB by 2050. The optimal long-term strategy would be a combination of serial mass campaigns in adults, coupled with universal newborn vaccination. Newborns are the only human population without prior mycobacterial exposure in TB endemic countries and we hypothesize that live attenuated mycobacterial vaccines will offer better protection to this naïve population compared to adults.

The objective of this project is to demonstrate safety, immunogenicity and improved efficacy of the new live attenuated M. tuberculosis vaccine called MTBVAC in a Phase 3 efficacy trial in HIV-uninfected infants born to HIV-infected and HIV-uninfected mothers as compared to standard of care BCG vaccination. The proposal builds upon a group of TB vaccine development partners in Europe and sub-Saharan Africa established in a previous EDCTP-supported project. It creates an expanded consortium of clinical trial partners for the optimal implementation of a large infant efficacy trial of MTBVAC in high TB incidence settings. New capacity for efficacy trials in infants will be a valuable resource for the TB vaccine development community. The proposal will create a network of institutions in three TB endemic African countries with enhanced laboratory capacity to conduct TB vaccine immunology studies and to bio-bank samples to discover immune correlates of vaccine-mediated protection.

MTBVAC is a novel TB vaccine candidate based on an attenuated M. tuberculosis clinical isolate of the Euro-American lineage. Attenuation is based on two independent, stable genetic deletions of the genes phoP and fadD26 coding for two major virulence factors, the transcription factor PhoP and the cell-wall lipids PDIM, respectively. The hypothesis is that MTBVAC will provide improved protection, as individuals latently infected with live M.tuberculosis have an 80% lower chance of developing TB, and as MTBVAC contains most of the genes deleted from BCG and presents a wider collection of antigens to the host immune system. Preclinical studies in different animal models indicated that MTBVAC is safe and is able to induce an improved protection compared to BCG.

Phase 1 studies showed that MTBVAC was safe and immunogenic in naïve adults and newborns, and evoked an immune response that exceeded the magnitude of BCG-induced immune responses. Larger dose-defining Phase 2a studies in newborns and in adults at extended dose-ranges to confirm these findings will be finalised in early 2021, and allow selection of a vaccine dose to progress into the proposed multi-centre efficacy trial in infants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female newborns within seven days of birth.
* Written informed maternal consent, including permission to access maternal antenatal, postnatal, and infant medical records.
* Infant participants and their caregivers available for trial follow-up and display the willingness and capacity to comply with trial procedures.
* Newborns must be in good general health during pregnancy and delivery, as assessed by medical history and targeted physical examination.
* Birth weight ≥ 2450 grams.
* Apgar score at 5 minutes ≥ 7.
* A maternal HIV test result (rapid test, enzyme-linked immunosorbent assay (ELISA), or Polymerase chain reaction (PCR)) taken within 30 days of delivery, or within seven days post-partum must be available and documented if HIV uninfected. If the mother is HIV infected, then she must be on antiretroviral (ARV) therapy as per in-country guidelines with a viral load of <50 copies/mL (within six months of labour).
* Estimated gestational age ≥ 37 weeks.
* Mother has not participated in a clinical trial within three months prior to the infant's birth.
* Mother has never participated in a TB vaccine trial before.
* Infant may not participate in any other clinical trials.

Exclusion Criteria:

Receipt of BCG vaccination prior to enrolment.

* Significant antenatal, intrapartum, or postpartum complications that may affect the health of the newborn.
* Skin condition, bruising or birth mark at the intended injection site.
* Maternal HIV test (rapid test, ELISA, or PCR) result not available.
* HIV exposed Newborn's HIV PCR result positive or not available.
* Maternal history of TB during pregnancy.
* History of close/household contact with a TB patient, antenatal or postnatal, whether maternal, other family member or another household member who has not yet completed TB treatment.
* Clinically suspected neonatal sepsis.
* Any severe congenital malformation.
* History or evidence of any systemic disease on examination, or any illness that in the opinion of the Investigator may interfere with the evaluation of the safety and immunogenicity of the vaccine. Neonatal jaundice not considered clinically significant is not an exclusion.

Ages: 5 Minutes to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7120 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
To demonstrate efficacy in terms of incidence of MTBVAC against TB disease in healthy HU and HEU newborns compared to BCG | Minimum of 24 months to a maximum 80 months; or until study end in South Africa.
  Primary: Time from vaccination to diagnosis of first confirmed or unconfirmed TB disease, which might be right-censored due to loss to follow-up, death, or successful completion of the study without acquiring TB disease from day of vaccination. Secondary: Confirmed TB disease, which might be right-censored due to loss to follow-up, death, or successful completion of the study without acquiring TB from day of vaccination. Exploratory: i) Time from vaccination to diagnosis of first unconfirmed or unlikely TB disease, which might be right-censored due to loss to follow-up, death, or successful completion of the study without acquiring TB disease from day of vaccination. ii) Confirmed or unconfirmed TB, which might be right-censored due to loss to follow-up, death, or successful completion of the study without acquiring TB carried out with a washout period of 90 days after vaccination. iii) Confirmed TB disease; iv) Unconfirmed or unlikely TB disease (ver ii for iii and iv).

SECONDARY OUTCOMES:
To assess the safety and reactogenicity of MTBVAC in healthy HU and HEU newborns compared to BCG. | Minimum of 24 months to a maximum 80 months; or until study end in South Africa.
  Incidence and severity of: Solicited AEs; Local solicited AEs (injection-site reactions): pain, erythema (redness), swelling, and induration (collected up to Day 10), and ulceration, drainage/discharge, and scarring (collected up to Day 56); Systemic solicited AEs: fever, irritability, vomiting, diarrhea, and skin rash (collected up to Day 10). Unsolicited AEs: MAAEs; Medically un-attended AEs. Solicited AEs with onset after Day 10: Local solicited AEs (injection-site reactions): pain, erythema (redness), swelling, and induration. Systemic solicited AEs: fever, irritability, vomiting, diarrhea, and skin rash. Solicited AEs with onset after Day 56: ulceration, drainage/discharge, and scarring; AESIs, SAEs

OTHER OUTCOMES:
Tertiary objective: To assess immunogenicity of MTBVAC in healthy HU and HEU newborns. | Minimum of 24 months to a maximum 80 months; or until study end in South Africa.
  • Frequencies and co-expression patterns of CD4 and CD8 T cells expressing IFNγ, TNF, IL-2, IL-17, and/or IL-22 induced by MTBVAC or BCG vaccination detected by WB-ICS after in vitro stimulation with MTBVAC, BCG, or a megapool of mycobacterial peptides.
Exploratory objective: To assess immunogenicity of MTBVAC in healthy HU and HEU newborns. | Minimum of 24 months to a maximum 80 months; or until study end in South Africa.
  Qualitative (positive or negative) and quantitative (TB Ag-Nil IFNγ concentration) QFT-Gold Plus assay results (QFT conversion will be defined as a positive test without a prior positive test; QFT reversion will be defined as a negative test following a positive test).
Exploratory objective: To biobank samples for (future) biomarker studies to identify immunological correlates of vaccine-induced protection and biomarkers of risk for TB disease | Minimum of 24 months to a maximum 80 months; or until study end in South Africa.
  • The following samples will be collected and biobanked for future studies to investigate the immune correlates of TB infection:
  * PBMC
  * Plasma
  * Paxgene The analyses will be described in a separate document.
Exploratory objective: To assess the non-specific effects of MTBVAC in healthy HU and HEU newborns compared to BCG. | Minimum of 24 months to a maximum 80 months; or until study end in South Africa.
  Primary
  • SAEs (hospitalization, death) due to non-TB infectious diseases classified as MedDRA SOC Infections and infestations occurring from Days 0 to 42.
  Secondary
  * MAAEs due to non-TB infectious diseases classified as MedDRA SOC Infections and infestations occurring from Days 0 to 42.
  * SAEs (hospitalization, death) due to non-TB infectious diseases classified as MedDRA SOC Infections and infestations occurring from Day 42 to EoSe.
  * MAAEs due to non-TB infectious diseases classified as MedDRA SOC Infections and infestations occurring from Day 42 to EoSe.
  * SAEs (hospitalization, death) occurring from Days 0 to 42 (or receipt of another vaccine type).
  * MAAEs occurring from Days 0 to 42 (or receipt of another vaccine type).
  * SAEs (hospitalization, death) from Day 42 to EoSe.
  * MAAEs from Day 42 to EoSe.
Exploratory objective: To assess TB case definitions determined by study-specific TB investigations compared to non-study solicited TB investigations in South Africa | Minimum of 24 months to a maximum 80 months; or until study end in South Africa.
  * Time from vaccination to diagnosis of first confirmed or unconfirmed TB disease, which might be right-censored due to loss to follow-up, death, or successful completion of the study without acquiring TB disease from the day of the vaccination.
  * Time from vaccination to diagnosis of first confirmed TB disease, which might be right-censored due to loss to follow-up, death, or successful completion of the study without acquiring TB disease from the day of the vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hatherill, Principal Investigator — University of Cape Town, Faculty of Health Sciences
Locations (1):
- South African Tuberculosis Initiative, Brewelskloof Hospital, Worcester, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tameris M, Mearns H, Penn-Nicholson A, Gregg Y, Bilek N, Mabwe S, Geldenhuys H, Shenje J, Luabeya AKK, Murillo I, Doce J, Aguilo N, Marinova D, Puentes E, Rodriguez E, Gonzalo-Asensio J, Fritzell B, Thole J, Martin C, Scriba TJ, Hatherill M; MTBVAC Clinical Trial Team. Live-attenuated Mycobacterium tuberculosis vaccine MTBVAC versus BCG in adults and neonates: a randomised controlled, double-blind dose-escalation trial. Lancet Respir Med. 2019 Sep;7(9):757-770. doi: 10.1016/S2213-2600(19)30251-6. Epub 2019 Aug 12. PMID 31416768
- [Background] Spertini F, Audran R, Chakour R, Karoui O, Steiner-Monard V, Thierry AC, Mayor CE, Rettby N, Jaton K, Vallotton L, Lazor-Blanchet C, Doce J, Puentes E, Marinova D, Aguilo N, Martin C. Safety of human immunisation with a live-attenuated Mycobacterium tuberculosis vaccine: a randomised, double-blind, controlled phase I trial. Lancet Respir Med. 2015 Dec;3(12):953-62. doi: 10.1016/S2213-2600(15)00435-X. Epub 2015 Nov 17. PMID 26598141
- [Background] Arbues A, Aguilo JI, Gonzalo-Asensio J, Marinova D, Uranga S, Puentes E, Fernandez C, Parra A, Cardona PJ, Vilaplana C, Ausina V, Williams A, Clark S, Malaga W, Guilhot C, Gicquel B, Martin C. Construction, characterization and preclinical evaluation of MTBVAC, the first live-attenuated M. tuberculosis-based vaccine to enter clinical trials. Vaccine. 2013 Oct 1;31(42):4867-73. doi: 10.1016/j.vaccine.2013.07.051. Epub 2013 Aug 17. PMID 23965219
- [Background] Aguilo N, Gonzalo-Asensio J, Alvarez-Arguedas S, Marinova D, Gomez AB, Uranga S, Spallek R, Singh M, Audran R, Spertini F, Martin C. Reactogenicity to major tuberculosis antigens absent in BCG is linked to improved protection against Mycobacterium tuberculosis. Nat Commun. 2017 Jul 14;8:16085. doi: 10.1038/ncomms16085. PMID 28706226
- [Background] Andrews JR, Noubary F, Walensky RP, Cerda R, Losina E, Horsburgh CR. Risk of progression to active tuberculosis following reinfection with Mycobacterium tuberculosis. Clin Infect Dis. 2012 Mar;54(6):784-91. doi: 10.1093/cid/cir951. Epub 2012 Jan 19. PMID 22267721
- [Background] Camacho LR, Ensergueix D, Perez E, Gicquel B, Guilhot C. Identification of a virulence gene cluster of Mycobacterium tuberculosis by signature-tagged transposon mutagenesis. Mol Microbiol. 1999 Oct;34(2):257-67. doi: 10.1046/j.1365-2958.1999.01593.x. PMID 10564470
- [Background] Copin R, Coscolla M, Efstathiadis E, Gagneux S, Ernst JD. Impact of in vitro evolution on antigenic diversity of Mycobacterium bovis bacillus Calmette-Guerin (BCG). Vaccine. 2014 Oct 14;32(45):5998-6004. doi: 10.1016/j.vaccine.2014.07.113. Epub 2014 Sep 6. PMID 25211768
- [Background] Gonzalo-Asensio J, Marinova D, Martin C, Aguilo N. MTBVAC: Attenuating the Human Pathogen of Tuberculosis (TB) Toward a Promising Vaccine against the TB Epidemic. Front Immunol. 2017 Dec 15;8:1803. doi: 10.3389/fimmu.2017.01803. eCollection 2017. PMID 29326700
- [Background] Gonzalo-Asensio J, Mostowy S, Harders-Westerveen J, Huygen K, Hernandez-Pando R, Thole J, Behr M, Gicquel B, Martin C. PhoP: a missing piece in the intricate puzzle of Mycobacterium tuberculosis virulence. PLoS One. 2008;3(10):e3496. doi: 10.1371/journal.pone.0003496. Epub 2008 Oct 23. PMID 18946503
- [Background] Graham SM, Ahmed T, Amanullah F, Browning R, Cardenas V, Casenghi M, Cuevas LE, Gale M, Gie RP, Grzemska M, Handelsman E, Hatherill M, Hesseling AC, Jean-Philippe P, Kampmann B, Kabra SK, Lienhardt C, Lighter-Fisher J, Madhi S, Makhene M, Marais BJ, McNeeley DF, Menzies H, Mitchell C, Modi S, Mofenson L, Musoke P, Nachman S, Powell C, Rigaud M, Rouzier V, Starke JR, Swaminathan S, Wingfield C. Evaluation of tuberculosis diagnostics in children: 1. Proposed clinical case definitions for classification of intrathoracic tuberculosis disease. Consensus from an expert panel. J Infect Dis. 2012 May 15;205 Suppl 2(Suppl 2):S199-208. doi: 10.1093/infdis/jis008. Epub 2012 Mar 22. PMID 22448023
- [Background] Kamath AT, Fruth U, Brennan MJ, Dobbelaer R, Hubrechts P, Ho MM, Mayner RE, Thole J, Walker KB, Liu M, Lambert PH; AERAS Global TB Vaccine Foundation; World Health Organization. New live mycobacterial vaccines: the Geneva consensus on essential steps towards clinical development. Vaccine. 2005 May 31;23(29):3753-61. doi: 10.1016/j.vaccine.2005.03.001. Epub 2005 Mar 24. PMID 15893612
- [Background] Knight GM, Griffiths UK, Sumner T, Laurence YV, Gheorghe A, Vassall A, Glaziou P, White RG. Impact and cost-effectiveness of new tuberculosis vaccines in low- and middle-income countries. Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15520-5. doi: 10.1073/pnas.1404386111. Epub 2014 Oct 6. PMID 25288770
- [Background] Marais S, Thwaites G, Schoeman JF, Torok ME, Misra UK, Prasad K, Donald PR, Wilkinson RJ, Marais BJ. Tuberculous meningitis: a uniform case definition for use in clinical research. Lancet Infect Dis. 2010 Nov;10(11):803-12. doi: 10.1016/S1473-3099(10)70138-9. Epub 2010 Sep 6. PMID 20822958
- [Background] Scriba TJ, Kaufmann SH, Henri Lambert P, Sanicas M, Martin C, Neyrolles O. Vaccination Against Tuberculosis With Whole-Cell Mycobacterial Vaccines. J Infect Dis. 2016 Sep 1;214(5):659-64. doi: 10.1093/infdis/jiw228. Epub 2016 May 30. PMID 27247343
- [Background] Stucki D, Brites D, Jeljeli L, Coscolla M, Liu Q, Trauner A, Fenner L, Rutaihwa L, Borrell S, Luo T, Gao Q, Kato-Maeda M, Ballif M, Egger M, Macedo R, Mardassi H, Moreno M, Tudo Vilanova G, Fyfe J, Globan M, Thomas J, Jamieson F, Guthrie JL, Asante-Poku A, Yeboah-Manu D, Wampande E, Ssengooba W, Joloba M, Henry Boom W, Basu I, Bower J, Saraiva M, Vaconcellos SEG, Suffys P, Koch A, Wilkinson R, Gail-Bekker L, Malla B, Ley SD, Beck HP, de Jong BC, Toit K, Sanchez-Padilla E, Bonnet M, Gil-Brusola A, Frank M, Penlap Beng VN, Eisenach K, Alani I, Wangui Ndung'u P, Revathi G, Gehre F, Akter S, Ntoumi F, Stewart-Isherwood L, Ntinginya NE, Rachow A, Hoelscher M, Cirillo DM, Skenders G, Hoffner S, Bakonyte D, Stakenas P, Diel R, Crudu V, Moldovan O, Al-Hajoj S, Otero L, Barletta F, Jane Carter E, Diero L, Supply P, Comas I, Niemann S, Gagneux S. Mycobacterium tuberculosis lineage 4 comprises globally distributed and geographically restricted sublineages. Nat Genet. 2016 Dec;48(12):1535-1543. doi: 10.1038/ng.3704. Epub 2016 Oct 31. PMID 27798628
- [Background] Tait DR, Hatherill M, Van Der Meeren O, Ginsberg AM, Van Brakel E, Salaun B, Scriba TJ, Akite EJ, Ayles HM, Bollaerts A, Demoitie MA, Diacon A, Evans TG, Gillard P, Hellstrom E, Innes JC, Lempicki M, Malahleha M, Martinson N, Mesia Vela D, Muyoyeta M, Nduba V, Pascal TG, Tameris M, Thienemann F, Wilkinson RJ, Roman F. Final Analysis of a Trial of M72/AS01E Vaccine to Prevent Tuberculosis. N Engl J Med. 2019 Dec 19;381(25):2429-2439. doi: 10.1056/NEJMoa1909953. Epub 2019 Oct 29. PMID 31661198
- [Background] Tameris MD, Hatherill M, Landry BS, Scriba TJ, Snowden MA, Lockhart S, Shea JE, McClain JB, Hussey GD, Hanekom WA, Mahomed H, McShane H; MVA85A 020 Trial Study Team. Safety and efficacy of MVA85A, a new tuberculosis vaccine, in infants previously vaccinated with BCG: a randomised, placebo-controlled phase 2b trial. Lancet. 2013 Mar 23;381(9871):1021-8. doi: 10.1016/S0140-6736(13)60177-4. PMID 23391465
- [Background] Walker KB, Brennan MJ, Ho MM, Eskola J, Thiry G, Sadoff J, Dobbelaer R, Grode L, Liu MA, Fruth U, Lambert PH. The second Geneva Consensus: Recommendations for novel live TB vaccines. Vaccine. 2010 Mar 8;28(11):2259-70. doi: 10.1016/j.vaccine.2009.12.083. Epub 2010 Jan 20. PMID 20074686
- [Background] White AD, Sibley L, Sarfas C, Morrison A, Gullick J, Clark S, Gleeson F, McIntyre A, Arlehamn CL, Sette A, Salguero FJ, Rayner E, Rodriguez E, Puentes E, Laddy D, Williams A, Dennis M, Martin C, Sharpe S. MTBVAC vaccination protects rhesus macaques against aerosol challenge with M. tuberculosis and induces immune signatures analogous to those observed in clinical studies. NPJ Vaccines. 2021 Jan 4;6(1):4. doi: 10.1038/s41541-020-00262-8. PMID 33397991
- [Background] Whitehead J. Overrunning and underrunning in sequential clinical trials. Control Clin Trials. 1992 Apr;13(2):106-21. doi: 10.1016/0197-2456(92)90017-t. PMID 1316826
- [Derived] Giersing B, Mo AX, Hwang A, Baqar S, Earle K, Ford A, Deal C, Dull P, Friede M, Hall BF. Meeting summary: Global vaccine and immunization research forum, 2023. Vaccine. 2025 Feb 6;46:126686. doi: 10.1016/j.vaccine.2024.126686. Epub 2025 Jan 5. PMID 39752894
- See also: WHO, Global Tuberculosis Report 2022. [Online] https://www.who.int/publications /i/item/9789240061729 [accessed on 27 June 2023]. — https://www.who.int/publications/i/item/9789240061729
- See also: WHO preferred products characteristics for TB vaccines 2018. [Online] https://apps.who.int/iris/ bitstream/handle/10665/273089/ WHO-IVB-18.06-eng.pdf?ua=1 [accessed on 05 May 2021]. — https://cdn.who.int/media/docs/default-source/immunization/product-and-delivery-research/framework_working_document_july_2023.pdf?sfvrsn=224b6151_3&download=true
- See also: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017. [Online] https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables [Accessed on 05 May 2021]. — https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf